CLINICAL TRIAL: NCT06181604
Title: Multicenter Symphony IL-6 Monitoring Sepsis ICU Pilot Study
Brief Title: Multicenter Symphony IL-6 Monitoring Sepsis ICU Study
Acronym: SYMON
Status: Completed | Type: Observational
Sponsor: Bluejay Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CES-0007
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Sepsis; Septic Shock
Keywords: Interleukin-6; IL-6; Risk Stratification; Infections; Toxemia; Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes; Sepsis; Septic Shock; Shock
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections; Toxemia; Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes; Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this study is to establish an IL-6 concentration cutoff and optimal time point(s) for using Symphony IL-6 that predict 28-day mortality in patients who are admitted or are intended to be admitted to the intensive care unit (ICU) diagnosed with sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥22 years of age)
* Diagnosis of sepsis or septic shock based on: the Third International Consensus Definitions (Sepsis-3 criteria) defined as at least one of the following criteria as determined by a treating physician or study physician investigator.
* Admitted or intended to be admitted to the ICU
* At least 0.4ml plasma drawn and available for collection (or is anticipated to be able to be drawn and available) within 12 hours of the earliest diagnosis of sepsis or septic shock.

Exclusion Criteria:

* Prisoners or imprisonment at time of enrollment
* Prior enrollment into this study
* Informed consent as approved by IRB is unable to be obtained.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with sepsis or septic shock, in accordance with the Sepsis-3 criteria, admitted or intended to be admitted to the ICU.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
28-day all-cause mortality | Within 28 days after inclusion
  Participants will be followed up for 28 days for all-cause mortality

SECONDARY OUTCOMES:
In-hospital mortality up to 28 days | Within 28 days after inclusion
  Participants will be followed up for 28 days for in-hospital mortality

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University of St. Louis, St Louis, Missouri
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - The Ohio State University/Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Healthcare, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No